CLINICAL TRIAL: NCT05125289
Title: Gender Based Comparison of Graston Technique, Active Release Technique and PNF Stretching on Hamstring Flexibility in Patients With Knee Osteoarthritis
Brief Title: Comparison of Soft Tissue Techniques on Hamstring Flexibility Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Ume habiba
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Knee Osteoarthritis
Keywords: Active release technique; Graston technique; Knee Osteoarthritis; PNF stretching; Hamstring tightness
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental intervention group 1 (Experimental): Graston technique group
  Interventions: Other: Graston technique group
- Experimental :interventional group II (Experimental): Active release technique group
  Interventions: Other: Active release technique group
- experimental group III (Experimental): Proprioceptive Neuromuscular Facilitation stretching group
  Interventions: Other: Proprioceptive Neuromuscular Facilitation stretching group

INTERVENTIONS:
Other: Graston technique group — Moist hot pack (10 minutes) Isometric quadriceps exercises (10 repetitions) Straight leg raise (10 repetitions) Graston technique steps 6 long strokes by the GT1 instrument on the hamstring muscle longitudinally. The Graston technique duration will be 5 minutes
  Arms: experimental intervention group 1
Other: Active release technique group — * Moist hot pack (10 minutes)
  * Isometric quadriceps exercises (10 repetitions)
  * Straight leg raise (10 repetitions)
  ART steps:
  * Subject lies on the plinth in prone or in side lying position with the dominant side facing upwards.
  * Gentle tension is applied to the hamstring muscle along the entire length while stretching the leg in prone lying or side lying positions, depending on the level of pain and tightness of muscle (5 repetitions at 5 seconds interval).
  * Gentle tension is also applied at the origin and insertion of the hamstring muscle until the patient feels full release.
  Arms: Experimental :interventional group II
Other: Proprioceptive Neuromuscular Facilitation stretching group — * Moist hot pack (10 minutes)
  * Isometric quadriceps exercises (10 repetitions)
  * Straight leg raise (10 repetitions)
  PNF technique steps:
  * The subject is in supine position with his non-dominant leg strapped down the table while the dominant leg rests on the therapist right shoulder.
  * The therapist stretches the hamstring muscle until the subject first reports a mild stretch sensation; held for 7 sec by passively flexing the hip with knee fully extended, allowing no hip rotation.
  * Next, the subject isometrically contracts the hamstring muscle for 3 sec and then relax for 5 sec.
  * This sequence is repeated 5 times at a 20 second interval.
  Arms: experimental group III

SUMMARY:
The aim of this research is to compare the effects of Graston Technique, active release technique and PNF stretching on hamstring flexibility in Patients with Knee Osteoarthritis. Randomized controlled trials done at Riphah International University, Islamabad.. The sample size was 45. The subjects were divided in three groups, 15 subjects in Graston Technique group, 15 subjects in active release technique group and 15 in PNF stretching group. Study duration was of 6 months. Sampling technique applied was non probability purposive sampling technique. Male and female patients greater than 30 years of age, with unilateral or bilateral OA of grade 1 and 2 in Kellegren and Lawrence criteria for knee OA, having UL/BL hamstring tightness, Pain > 3 on NPRS, ROM > 200 from AKE test were included.

Tools used in the study are NPRS, AKE test by goniometer, Lower extremity functional index (LEFI) and WOMAC.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis, affecting an estimated 302 million people worldwide. It is expected that ten percent males and 18 percent females have knee or hip OA. It ranks as the fifth highest cause of years lost to disability in the whole population in high-income countries, and the ninth highest cause in low- and middle-income countries. In older people, OA is the utmost devastating musculoskeletal syndrome.

It is a long-term chronic disease characterized by the destruction of articular cartilage and underlying bone. The degeneration occurs due to disarrangement in the usual process of repair of a joint. When the process breaks the synchronicity, there is slow deterioration of the articular cartilage. As a result, the biomechanical influences on the joints are also changed due to loss of normal joint line of gravity. This ultimately leads toward symptomatic changes which are a focal loss of the cartilage covering the articular ends; loss of normal joint space requires for smooth grating, osteophyte formation in joint, and remoulding of bone on peripheral areas and along the articular sides. Signs and symptoms are pain, a restricted range of joint movement, reduced muscle strength, restricted activities of daily living (ADLs) and instrumental activities of daily living (IADLS), and reduced quality of life.

Exercise, weight loss in patients with knee and/or hip OA who are overweight or obese, self-efficacy and self-management programs, tai chi, cane use, hand orthoses for first carpometacarpal (CMC) joint OA, tibiofemoral bracing for tibiofemoral knee OA, topical nonsteroidal anti-inflammatory drugs (NSAIDs) for knee OA, oral NSAIDs, and intraarticular glucocorticoid injections for knee OA are strongly recommended for treatment purposes. One major problem for patients with knee OA is poor hamstring flexibility. The stretching of the hamstring is a necessary intervention in the management of the OA knee. Although research and clinical experience has shown that treatment of hamstring flexibility is important, there is no widely acceptable form of treatment that is agreed upon to successfully improve flexibility of hamstrings.

Instrument assisted soft tissue mobilization (IASTM) using Graston technique is a popular treatment for myofascial restriction. The IASTM treatment is thought to stimulate connective tissue remodeling through resorption of excessive fibrosis, along with inducing repair and regeneration of collagen secondary to fibroblast recruitment. In turn, this will result in the release and breakdown of scar tissue, adhesions, and fascial restrictions.

Active release technique (ART) is also a technique that involves breaking down adhesions and scar tissue which cause pain and dysfunctions. It involves a clinician using their thumbs or fingers to apply deep tension to a trigger point while the involved tissue is moved from a shortened to lengthened position both actively by the patient and passively by the clinician.

Proprioceptive Neuromuscular Facilitation (PNF) stretching technique is another technique utilized to improve muscle elasticity. This technique is specifically designed to stimulate mechanoreceptors and significant effect of static as well as PNF stretching on clinical symptoms of knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 30years. Both male & female. Uni/bilateral OA. Grade I or II OA. Uni/bilateral hamstring tightness ranging between 40 to 70 degrees of a straight leg raise.

Exclusion Criteria:

* Hamstring injury and strains within 2 months. Any skin infections History of any lower limb surgeries within last 6 months. Lumber disc herniation. Lower limb neurological compromise.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
WOMAC | 4th week
  WOMAC was used for evaluating Osteoarthritis patients. The WOMAC OA index included 24 questions and three sections that questioned pain, stiffness, and physical function. The scale included five pain-related questions, two stiffness-related questions, and 17 physical function- related questions. The maximum scores were 20 for the pain subgroup, eight for the stiffness subgroup and 68 for the physical function subgroup. High scores indicated that the patient had worse symptoms in the relevant group.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS) | 4th week
  NPRS was used for one-dimensional pain measurement It was an 11-item scale in which respondents selected the whole number from 0 to 10 to best describe their pain intensity in the last 24 hours. 0 represented no pain and 10 represented the worst possible pain experienced by the respondent. It had a reliability of 0.96 in literate and 0.95 in illiterate patients and had 0.86 - 0.95 validity.
Active Knee Extension Test | 4th week
  The AKET measured hamstring muscle length. In the AKET, the patient actively extended the knee until reaching maximal stretch of the hamstring while the ipsilateral hip was kept at a fixed angle, usually 90 or 120 degrees of flexion.
Lower extremity functional index | 4th week
  The lower extremity functional scale is a well-known and validated patient-rated outcome measure (PROM) that was used to measure lower extremity function. The score consisted of 20 questions, which were subdivided into 4 groups. These groups consisted of activities with increasing physical demands. Questions on activity varied from walking between rooms to running on uneven ground.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, MSPT-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No